CLINICAL TRIAL: NCT01831804
Title: Phase I Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of Topical GSK1278863 in Healthy Volunteers and Diabetic Patients, and Repeat Doses of GSK1278863 in Diabetic Patients for the Treatment of Diabetic Foot Ulcer
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Single and Repeated Doses of Topical GSK1278863
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 115760
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-06

CONDITIONS: Wound Healing
Keywords: diabetic foot ulcer; pharmacodynamics; pharmacokinetics; ischemic
MeSH Terms: conditions — Diabetic Foot; Ischemia | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 Part A (Experimental): Healthy subjects in this arm will receive single applications of GSK1278863 or placebo (with 6:2 ratio) on intact skin in two escalating dosing periods each separated by 10 days. The first application will be with a single dose of 0.3 mg and second application will be single dose of 3 mg.
  Interventions: Drug: GSK1278863; Drug: Placebo
- Cohort 2 Part A (Experimental): Subjects with diabetic foot ulcer (DFU) will receive a single application of GSK1278863 or placebo (with 6:2 ratio) in two dosing periods separated by 10 days. The first application will be made on intact skin and second application directly on DFU. Dose will be based on wound area and review from previous cohort data.
  Interventions: Drug: GSK1278863; Drug: Placebo
- Cohort 3 Part A (Experimental): Subjects with DFU will receive single application of GSK1278863 or placebo directly on DFU. Dose will be based on wound area and review from previous cohort data.
  Interventions: Drug: GSK1278863; Drug: Placebo
- Cohort 4 Part A (Experimental): Subjects with DFU will receive a single application of GSK1278863 or placebo (with 6:2 ratio) in two dosing periods separated by 10 days. The first application will be made on DFU and second application on intact skin. Dose will be based on wound area and review from previous cohort data.
  Interventions: Drug: GSK1278863; Drug: Placebo
- Cohort 5 Part B (Experimental): Subjects with DFU will receive Standard of care (SOC) up to 15 days and then will be randomized to one of the three arms: GSK1278863 + SOC, or SOC only, or placebo + SOC with ratio of 12:2:2. Doses for the cohorts in Part B will be determined from safety, tolerability and PK data from Part A. subjects will first be given a single application of GSK1278863 or placebo at the dose chosen for that cohort, followed by a 7-day washout period, and then repeat applications for 14 days, starting on Day 8.
  Interventions: Drug: GSK1278863; Drug: Placebo
- Cohort 6 Part B (Experimental): Subjects with DFU will receive Standard of care (SOC) up to 15 days and then will be randomized to one of the three arms: GSK1278863 + SOC, or SOC only, or placebo + SOC with ratio of 12:2:2. Doses for the cohorts in Part B will be determined from safety, tolerability and PK data from Part A. subjects will first be given a single application of GSK1278863 or placebo at the dose chosen for that cohort, followed by a 7-day washout period, and then repeat applications for 14 days, starting on Day 8.
  Interventions: Drug: GSK1278863; Drug: Placebo
- Cohort 7 Part B (Experimental): Subjects with DFU will receive Standard of care (SOC) up to 15 days and then will be randomized to one of the three arms: GSK1278863 + SOC, or SOC only, or placebo + SOC with ratio of 12:2:2. Doses for the cohorts in Part B will be determined from safety, tolerability and PK data from Part A. subjects will first be given a single application of GSK1278863 or placebo at the dose chosen for that cohort, followed by a 7-day washout period, and then repeat applications for 14 days, starting on Day 8.
  Interventions: Drug: GSK1278863; Drug: Placebo

INTERVENTIONS:
Drug: GSK1278863 — White to off-white smooth ointment with unit dose strength of 0.05%w/w, 0.1%w/w, 0.5%w/w, 1.0%w/w for topical application as single or repeat doses.
Drug: Placebo — White to off-white smooth ointment for topical application as single or repeat doses.

SUMMARY:
This is a randomized, placebo-controlled, single-blind (subjects and investigators will be blinded, GSK internal personnel will not be blinded), parallel-group, two part (Part A, Part B) trial in healthy volunteers and subjects with diabetic foot ulcers. Part A is designed to evaluate single applications of GSK1278863 in one cohort of healthy volunteers (intact skin) and approximately 3 cohorts of diabetic subjects. Part B is designed to evaluate first single, and then repeat applications of GSK1278863 in diabetics, both in the clinic and by subjects at home. Part B will include approximately 3 cohorts in which the concentration of drug applied will be determined by pharmacokinetic data from Part A and earlier cohorts in Part B.

ELIGIBILITY:
Inclusion Criteria - Healthy Volunteers (Part A Cohort 1)

* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* [Single] corrected QT interval (QTc) < 450 millisecond (msec).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and electrocardiogram (ECGs). A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with hemoglobin (Hb) values higher than ULN the normal range should always be excluded from enrollment.
* Male or female between 18 and 90 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential (postmenopausal or pre-menopausal females with a documented tubal ligation or hysterectomy). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol.

Inclusion Criteria - DFU Subjects must meet healthy volunteer inclusion criteria and the following

* Diagnosed with Type I or Type II diabetes mellitus.
* Glycosylated haemoglobin (HbA1c) <=12%.
* QTc < 480 msec in subjects with bundle branch block.
* Lower extremity diabetic foot ulcer of 30 to 364 days' duration.
* DFU between 1 centimeter squared (cm ^2) and 20 cm^2 at screening.
* Presence of at least one DFU that meets all of the following criteria: (a). Ulcer has been diagnosed as a full-thickness, neuropathic DFU and is located at or distal to the malleolus (excluding ulcers between the toes but including those of the heel). (b). There is a minimum 2 cm margin between the qualifying study ulcer and any other ulcers on the specified foot. (c). Ulcer size (area) >=1 cm^2 and <=12 cm^2 (post-debridement at time of randomization). (d). Wagner Grade 1. (e). Depth <=5 millimeter (mm) with no capsule, tendon or bone exposed and no tunneling, undermining, or sinus tracts. Note: If the subject has more than one qualifying DFU, the ulcer designated as the study ulcer will be at the discretion of the Investigator. Non-study ulcers being treated during the course of the study will be treated with moist wound therapy Standard of Care (SOC) identified under this study.
* Adequate vascular perfusion of the affected limb within 30 days of screening, as defined by at least one of the following: (a) Transcutaneous oxygen partial pressure (TcPO2) >35 millimeter of mercury (mmHg). (b) Ankle-Brachial Index (ABI) >=0.6 and <=1.2, confirmed by TcPO2 >35 mmHg. (c) Toe pressure (plethysmography) >50 mmHg. (d) Doppler ultrasound (biphasic or triphasic waveforms) consistent with adequate blood flow to the affected extremity, as determined by SOC.

Exclusion Criteria - Healthy Volunteers (Part A Cohort 1)

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of malignancy within 5 years of Screening or those with a strong family history of cancer (e.g., familial cancer disorders), with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated.
* A history of drug or alcohol abuse, or a history of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 mililiter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* A positive test for human immunodeficiency virus (HIV) antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives (whichever is longer).
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.
* Pregnant females as determined by positive urine human chorionic gonadotropin test at screening or prior to dosing.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated. Exclusion Criteria - DFU Subjects

Healthy volunteer exclusions apply to DFU subjects in addition to the following:

* Subjects with ulcers accompanied by infected cellulitis, osteomyelitis, or clinical signs or symptoms of infection, Gangrene on any part of affected limb, Active Charcot's foot on the study limb, Planned vascular surgery, angioplasty or thrombolysis, Ulcers involving exposure of tendon, bone, or joint capsule (It is acceptable to have ulcers extending through the dermis and into subcutaneous tissue with presence of granulation tissue), Ulcers due to non-diabetic etiology.
* Any unstable vascular syndromes (such as transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, acute myocardial infarction (MI) or acute coronary syndrome event (ACS) and/or any major changes (per investigator's judgment) to related medications within 6 months prior to randomization.
* History or malignancy within 5 years of screening or those with a strong family history of cancer (e.g. familial cancer disorders), with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated.
* Other clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, hematological, or metabolic disease that is, in the opinion of the Investigator or the GSK Medical Monitor, not stabilized or may otherwise impact the results of the study.
* Patients with active treatment for retinal neovascularization (e.g., diabetic proliferative retinopathy or age related macular degeneration) within 6 months of randomization.
* Patients undergoing hemodialysis.
* History of venous thrombosis defined as deep vein thrombosis, pulmonary embolism or other venous thrombotic condition within 1 year prior to screening.
* Active peptic, duodenal, or esophageal ulcer disease or any gastrointestinal bleeding, within 1 year prior to screening.
* Subjects with a platelet count <100,000/mm^3 at screening.
* Subjects with an International Normalized Ratio (INR) >1.5 at screening.
* Subjects with a hemoglobin level above the gender-specific upper limit of normal at screening.
* Subjects with a history of non-traumatic joint inflammation (with the exception of inflammation due to osteoarthritis).
* Patients with known pulmonary hypertension.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-06-17 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, Castro Valley, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=SCD117226

REFERENCES:
- [Background] Olson E, Mahar KM, Morgan L, Fillmore C, Holland C, Lavery L. Randomized Phase I Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Topical Daprodustat in Healthy Volunteers and in Patients With Diabetic Foot Ulcers. Clin Pharmacol Drug Dev. 2019 Aug;8(6):765-778. doi: 10.1002/cpdd.654. Epub 2019 Feb 5. PMID 30720931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo-controlled, single-blind, parallel-group, two part (Part A and Part B) study in healthy volunteers (HVT) and participants with diabetic foot ulcer (DFU).
Pre-assignment Details: A total of 65 par. were randomized, however 2 par. did not receive study treatment and were excluded from analysis. All data tables reflect the total of treated par. (63).
Groups:
- Placebo HVT (Cohort 1): Cohort 1 comprised of healthy participants. Participants were administered a single dose of placebo on intact skin during two dosing periods. There was a wash out period of at least 10 days between the two periods.
- Placebo DFU SD (Cohort 2, 3, 4): Cohorts 2, 3 and 4 consisted of participants with DFU. Participants were administered a single dose of placebo in one (Cohort 3) or two (Cohort 2 and 4) dosing periods. There was a wash out period of at least 10 days between periods.
- A/B (Cohort 1): Healthy participants were enrolled. Participants were administered a single dose of treatment A=0.3 milligram (mg) GSK1278863 on intact skin in Period 1 and a single dose of treatment B=3 mg GSK1278863 on intact skin in Period 2. There was a wash out period of 10 days between the two periods.
- C/C (Cohort 2): Participants with DFU were administered 0.1 percent of 25 milligrams per square centimeter (mg/cm^2) GSK1278863 on intact skin in Period 1 followed by a wash-out period of at least 10 days. Participants were then administered a single dose of 0.1 percent of 25 mg/cm^2 on wounded skin in Period 2.
- D (Cohort 3): Participants with DFU were administered a single dose of 1 percent of 25 mg/cm^2 GSK1278863 on wounded skin.
- E/E (Cohort 4): A single dose of 1 percent of 100 mg/cm^2 GSK1278863 was applied directly to wounded skin in Period 1, followed by application of a single dose of 1 percent of 100 mg/cm^2 GSK1278863 to intact skin. There was a wash-out period of at least 10 days between the two dosing periods.
- Placebo DFU RD (Cohort 5): Participants with DFU received once daily placebo application directly to the wounded skin for 14 days along with standard of care therapy.
- R1r (Cohort 5): Participants with DFU received once daily application of 1 percent of 100 mg/cm^2 GSK1278863 to wounded skin for 14 days along with standard of care treatment.
- Sr (Cohort 5): Participants with DFU continued to receive daily application of standard of care wound treatment for 14 days.
Period: Overall Study
Arm/Group | Placebo HVT (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4) | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5)
Started | 4 | 3 | 9 | 5 | 5 | 3 | 4 | 26 | 4
Completed | 3 | 1 | 3 | 5 | 3 | 3 | 3 | 23 | 2
Not Completed | 1 | 2 | 6 | 0 | 2 | 0 | 1 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol defined stopping criteria | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Investigator discretion | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrew Consent | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo HVT (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4) | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5) | Total
Number analyzed (Participants) | 4 | 3 | 9 | 5 | 5 | 3 | 4 | 26 | 4 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (14.20) | 53.0 (8.72) | 44.4 (15.27) | 52.6 (5.90) | 59.2 (7.66) | 48.3 (11.93) | 50.0 (10.42) | 55.5 (6.13) | 55.5 (5.26) | 51.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 3 | 1 | 9
  Male | 3 | 3 | 6 | 5 | 5 | 3 | 3 | 23 | 3 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage (Her.) | 2 | 1 | 4 | 1 | 1 | 0 | 0 | 6 | 1 | 16
  Japanese/East Asian Her./South East Asian Her. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 2 | 2 | 5 | 4 | 4 | 3 | 4 | 19 | 3 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) Following Single Dose Administration (Part A)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; other important medical events; or is associated with liver injury and impaired liver function.
Time Frame: Up to a maximum of 75 days (Start of study treatment through final follow up 2 [28-32 days post last dose])
Population: All Subject Population comprised of all participants who received at least one dose of study drug (including GSK1278863, placebo and standard care).
Measure: Number; unit: Participants
Groups:
- C (Cohort 2): Participants with DFU were a single dose of 0.1 percent of 25 mg/cm^2 GSK1278863 on wounded skin.
- E (Cohort 4): Participants with DFU were administered a single dose of 1 percent of 100 mg/cm^2 GSK1278863 on wounded skin.
Arm/Group | Placebo HVT (Cohort 1) | A/B (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | C (Cohort 2) | D (Cohort 3) | E (Cohort 4)
Number analyzed (Participants) | 4 | 9 | 3 | 5 | 5 | 3
Participants
  AEs | 2 | 3 | 1 | 0 | 2 | 1
  SAEs | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With AEs and SAEs Following Repeat Dose Administration (Part B)
Description: as for outcome 1
Time Frame: Up to a maximum of 53 days (Start of study treatment through final follow up 2 [28-32 days post last dose])
Population: All Subject Population.
Measure: Number; unit: Participants
Arm/Group | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5)
Number analyzed (Participants) | 4 | 26 | 4
Participants
  AEs | 2 | 5 | 2
  SAEs | 1 | 0 | 1

3. Primary Outcome: Number of Participants With Clinically Significant 12-lead Electrocardiograms (ECGs) Measurement Following Single Dose Administrations (Part A)
Description: ECG measurements were taken with the participants in supine position for at least 5 minutes. The number of participants with clinically significant abnormal ECG measurement following single dose administration for worst case post-Baseline visit has been presented.
Time Frame: Up to a maximum of 75 days (Start of study treatment through final follow up 2 [28-32 days post last dose])
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Placebo HVT (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 4 | 3 | 9 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant 12-lead ECG Measurement Following Repeat Dose Administrations (Part B)
Description: as for outcome 3
Time Frame: Up to a maximum of 53 days (Start of study treatment through final follow up 2 [28-32 days post last dose])
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5)
Number analyzed (Participants) | 4 | 26 | 4
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Vital Sign Data Outside Clinical Concern Range Following Single Dose Administration (Part A)
Description: Vital sign measurements included systolic blood pressure (SBP) and diastolic blood pressure (DBP). Vital signs were measured after the participants rested in a supine or semi-supine position for 5 minutes prior to the procedure. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). When a high or low value was reported, all values are presented for that time point and parameter.
Time Frame: Day 1 (pre-dose and 48 hours) of Periods 1 and 2
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Placebo HVT (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 4 | 3 | 9 | 5 | 5 | 3
Participants
  DBP Period 2; Day 1; 48 hours; Low; n=4,1,0,5,0,3: number analyzed (Participants) | 4 | 1 | 0 | 5 | 0 | 3
  DBP Period 2; Day 1; 48 hours; Low; n=4,1,0,5,0,3 | 0 | 0 |  | 0 |  | 0
  DBP Period 2; Day 1; 48 hours; High; n=4,1,0,5,0,3: number analyzed (Participants) | 4 | 1 | 0 | 5 | 0 | 3
  DBP Period 2; Day 1; 48 hours; High; n=4,1,0,5,0,3 | 0 | 1 |  | 0 |  | 1
  SBP; Period 1; Day 1;pre-dose;Low;n=4,3,9,5,5,3 | 0 | 0 | 0 | 0 | 0 | 0
  SBP; Period 1; Day 1;pre-dose;High;n=4,3,9,5,5,3 | 0 | 0 | 0 | 2 | 1 | 0
  SBP; Period 1; Day 1;48 hours;Low;n=4,3,8,5,4,3: number analyzed (Participants) | 4 | 3 | 8 | 5 | 4 | 3
  SBP; Period 1; Day 1;48 hours;Low;n=4,3,8,5,4,3 | 0 | 0 | 0 | 0 | 0 | 0
  SBP; Period 1; Day 1;48 hours;High;n=4,3,8,5,4,3: number analyzed (Participants) | 4 | 3 | 8 | 5 | 4 | 3
  SBP; Period 1; Day 1;48 hours;High;n=4,3,8,5,4,3 | 0 | 0 | 0 | 2 | 0 | 1
  SBP; Period 2; Day 1;pre-dose;Low;n=4,2,0,5,0,3: number analyzed (Participants) | 4 | 2 | 0 | 5 | 0 | 3
  SBP; Period 2; Day 1;pre-dose;Low;n=4,2,0,5,0,3 | 0 | 0 |  | 0 |  | 0
  SBP; Period 2; Day 1;pre-dose;High;n=4,2,0,5,0,3: number analyzed (Participants) | 4 | 2 | 0 | 5 | 0 | 3
  SBP; Period 2; Day 1;pre-dose;High;n=4,2,0,5,0,3 | 0 | 0 |  | 1 |  | 0
  SBP; Period 2; Day 1;48 hours;Low;n=4,1,0,5,0,3: number analyzed (Participants) | 4 | 1 | 0 | 5 | 0 | 3
  SBP; Period 2; Day 1;48 hours;Low;n=4,1,0,5,0,3 | 0 | 0 |  | 0 |  | 0
  SBP; Period 2; Day 1;48 hours;High;n=4,1,0,5,0,3: number analyzed (Participants) | 4 | 1 | 0 | 5 | 0 | 3
  SBP; Period 2; Day 1;48 hours;High;n=4,1,0,5,0,3 | 0 | 0 |  | 1 |  | 1

6. Primary Outcome: Number of Participants With Vital Sign Data Outside Clinical Concern Range Following Repeat Dose Administration (Part B)
Description: as for outcome 5
Time Frame: Days 1 and 7 (pre-dose), Day 14 (24 hours)
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5)
Number analyzed (Participants) | 4 | 26 | 4
Participants
  DBP,Day 1,pre-dose,Low,n=4,26,4 | 0 | 0 | 0
  DBP,Day 1,pre-dose,High,n=4,26,4 | 0 | 1 | 0
  SBP,Day 1,pre-dose,Low, n=4,26,4 | 0 | 0 | 0
  SBP,Day 1,pre-dose,High, n=4,26,4 | 1 | 3 | 0
  SBP,Day 7,pre-dose,Low, n=4,25,4: number analyzed (Participants) | 4 | 25 | 4
  SBP,Day 7,pre-dose,Low, n=4,25,4 | 0 | 0 | 0
  SBP,Day 7,pre-dose,High, n=4,25,4: number analyzed (Participants) | 4 | 25 | 4
  SBP,Day 7,pre-dose,High, n=4,25,4 | 0 | 2 | 0
  SBP,Day 14,24 H,Low, n=3,22,1: number analyzed (Participants) | 3 | 22 | 1
  SBP,Day 14,24 H,Low, n=3,22,1 | 0 | 0 | 0
  SBP,Day 14,24 H,High, n=3,22,1: number analyzed (Participants) | 3 | 22 | 1
  SBP,Day 14,24 H,High, n=3,22,1 | 0 | 3 | 0

7. Primary Outcome: Number of Participants With Abnormal Nurse/Physician Observation (Part A)
Description: A brief physical assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen) were planned to be performed by qualified licensed, medical professional (i.e., physician, physician assistant, or nurse practitioner) but was not performed.Since data was not collected, no analysis was performed.
Time Frame: Up to a maximum of 75 days (Start of study treatment through final follow up 2 [28-32 days post last dose])
Population: All Subject Population
Arm/Group | Placebo HVT (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Abnormal Nurse/Physician Observation (Part B)
Description: A brief physical assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen) were planned to be performed by qualified licensed, medical professional (i.e., physician, physician assistant, or nurse practitioner) but was not performed. Since data was not collected, no analysis was performed.
Time Frame: Up to a maximum of 53 days (Start of study treatment through final follow up 2 [28-32 days post last dose])
Population: All Subject Population
Arm/Group | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5)
Number analyzed (Participants) | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Hematology Values Outside the Clinical Concern Range (Part A)
Description: Hematology parameters assessed were: platelet count, red blood cell count, white blood cell count, hemoglobin, reticulocyte count, hematocrit, absolute neutrophil count (ANC), monocytes, lymphocytes, eosinophils, basophils, mean corpuscular volume, mean corpuscular hemoglobin, and mean corpuscular hemoglobin concentration. When a high or low value was reported, all values are presented for that time point and parameter.
Time Frame: Day 1 (pre-dose)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Placebo HVT (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 4 | 3 | 9 | 5 | 5 | 3
Participants
  Total ANC,Day 1,pre-dose,Low | 0 | 1 | 1 | 0 | 0 | 0
  Total ANC,Day 1,pre-dose,High | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Hematology Data Outside the Clinical Concern Range (Part B)
Description: Hematology parameters assessed were: platelet count, red blood cell count, white blood cell count, hemoglobin, reticulocyte count, hematocrit, neutrophils, monocytes, lymphocytes, eosinophils, basophils, mean corpuscular volume, mean corpuscular hemoglobin, and mean corpuscular hemoglobin concentration. When a high or low value was reported, all values are presented for that time point and parameter.
Time Frame: Day 1 (pre-dose)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5)
Number analyzed (Participants) | 4 | 26 | 4
Participants
  Lymphocytes, Day 1,pre-dose,Low | 0 | 1 | 0
  Lymphocytes, Day 1,pre-dose,High | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Clinical Chemistry Values Outside the Clinical Concern Range (Part A)
Description: Chemistry parameters assessed were: Blood urea nitrogen (BUN), creatinine, fasting glucose, sodium, creatine phosphokinase (CPK), potassium, chloride, total carbon dioxide (CO2), calcium, glycosylated hemoglobin (HbA1C), Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Gamma glutamyltransferase (GGT), Alkaline phosphatase (ALP), High sensitivity C-reactive protein (hsCRP), total and direct bilirubin, uric acid, albumin and total protein. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). When a high or low value was reported, all values are presented for that time point and parameter.
Time Frame: Day 1 (pre-dose and 48 hours) in period 1; Day 1 (48 hours) in period 2
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Placebo HVT (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 4 | 3 | 9 | 5 | 5 | 3
Participants
  Glucose,Day1,P1,pre-dose,low,n=4,3,9,5,5,3 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose,Day1,P1,pre-dose,high,n=4,3,9,5,5,3 | 0 | 0 | 0 | 0 | 1 | 0
  Glucose,Day1,P1,48 H,low,n=4,3,8,5,4,3: number analyzed (Participants) | 4 | 3 | 8 | 5 | 4 | 3
  Glucose,Day1,P1,48 H,low,n=4,3,8,5,4,3 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose,Day1,P1,48 H,high,n=4,3,8,5,4,3: number analyzed (Participants) | 4 | 3 | 8 | 5 | 4 | 3
  Glucose,Day1,P1,48 H,high,n=4,3,8,5,4,3 | 0 | 0 | 0 | 0 | 0 | 1
  Glucose,Day1,P2,48 H,low,n=4,1,0,5,0,3: number analyzed (Participants) | 4 | 1 | 0 | 5 | 0 | 3
  Glucose,Day1,P2,48 H,low,n=4,1,0,5,0,3 | 0 | 0 |  | 0 |  | 0
  Glucose,Day1,P2,48 H,high,n=4,1,0,5,0,3: number analyzed (Participants) | 4 | 1 | 0 | 5 | 0 | 3
  Glucose,Day1,P2,48 H,high,n=4,1,0,5,0,3 | 0 | 0 |  | 1 |  | 2

12. Primary Outcome: Number of Participants With Clinical Chemistry Values Outside the Clinical Concern Range (Part B)
Description: as for outcome 11
Time Frame: Days 1 and 7 (pre-dose) and Day 14 (24 hours)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5)
Number analyzed (Participants) | 4 | 26 | 4
Participants
  Glucose,Day1,pre-dose,Low,n=4,26,4 | 0 | 0 | 0
  Glucose,Day1,pre-dose,High,n=4,26,4 | 0 | 5 | 1
  Glucose,Day7,pre-dose,Low,n=4,24,4: number analyzed (Participants) | 4 | 24 | 4
  Glucose,Day7,pre-dose,Low,n=4,24,4 | 0 | 0 | 0
  Glucose,Day7,pre-dose,High,n=4,24,4: number analyzed (Participants) | 4 | 24 | 4
  Glucose,Day7,pre-dose,High,n=4,24,4 | 0 | 7 | 2
  Glucose,Day14,24H,Low,n=3,23,2: number analyzed (Participants) | 3 | 23 | 2
  Glucose,Day14,24H,Low,n=3,23,2 | 0 | 0 | 0
  Glucose,Day14,24H,High,n=3,23,2: number analyzed (Participants) | 3 | 23 | 2
  Glucose,Day14,24H,High,n=3,23,2 | 2 | 9 | 0

13. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK1278863 (Part A)
Description: The pharmacokinetic (PK) parameters were calculated by standard non-compartmental analysis according to current working practices and using WinNonlin Version 5.2 or higher. All calculations of non-compartmental parameters were based on actual sampling times. Cmax could not be determined as data was below the limit of quantification.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72 hrs post-dose
Population: All participants from whom a PK sample had been obtained and analyzed were included in the PK Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 9 | 5 | 5 | 3
Nanograms per milliliter (ng/mL) | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

14. Primary Outcome: Cmax of GSK1278863 (Part B)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis according to current working practices and using WinNonlin Version 5.2 or higher. All calculations of non-compartmental parameters were based on actual sampling times. Cmax could not be determined as data was below the limit of quantification.
Time Frame: Pre-dose and 2 hrs on Day 1 and 7; pre-dose, 1, 2,4, 8, 12 and 24 hrs post-dose on Day 14
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | R1r (Cohort 5)
Number analyzed (Participants) | 26
ng/mL | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

15. Primary Outcome: Time of Occurrence of Cmax (Tmax) of GSK1278863 (Part A)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis according to current working practices and using WinNonlin Version 5.2 or higher. All calculations of non-compartmental parameters were based on actual sampling times. Tmax could not be determined as data was below the limit of quantification.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72hrs post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 9 | 5 | 5 | 3
Hour | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

16. Primary Outcome: Tmax of GSK1278863 (Part B)
Description: as for outcome 15
Time Frame: Pre-dose and 2 hrs on Day 1 and 7; pre-dose, 1, 2,4, 8, 12 and 24 hrs post-dose on Day 14
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | R1r (Cohort 5)
Number analyzed (Participants) | 26
Hour | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

17. Primary Outcome: Apparent Terminal Elimination Half-life (t1/2) of GSK1278863 (Part A)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis according to current working practices and using WinNonlin Version 5.2 or higher. All calculations of non-compartmental parameters were based on actual sampling times. t1/2 could not be determined as data was below the limit of quantification.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72hrs post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 9 | 5 | 5 | 3
Hour | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

18. Primary Outcome: t1/2 of GSK1278863 (Part B)
Description: as for outcome 17
Time Frame: Pre-dose and 2 hrs on Day 1 and 7; pre-dose, 1, 2,4, 8, 12 and 24 hrs post-dose on Day 14
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | R1r (Cohort 5)
Number analyzed (Participants) | 26
Hour | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

19. Primary Outcome: Lag Time Before Observation of Drug Concentrations in Sampled Matrix (Tlag) (Part A)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis according to current working practices and using WinNonlin Version 5.2 or higher. All calculations of non-compartmental parameters were based on actual sampling times. Tlag could not be determined as data was below the limit of quantification.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72hrs post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 9 | 5 | 5 | 3
Hour | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification..

20. Primary Outcome: Lag Time Before Observation of Drug Concentrations in Sampled Matrix (Tlag) (Part B)
Description: as for outcome 19
Time Frame: Pre-dose and 2 hrs on Day 1 and 7; pre-dose, 1, 2,4, 8, 12 and 24 hrs post-dose on Day 14
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | R1r (Cohort 5)
Number analyzed (Participants) | 26
Hour | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

21. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time [AUC(0-inf)] of GSK1278863 (Part A)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis according to current working practices and using WinNonlin Version 5.2 or higher. All calculations of non-compartmental parameters were based on actual sampling times. AUC (0-inf) could not be determined as data was below the limit of quantification.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72hrs post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: hour*nanograms/milliliter
Arm/Group | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 9 | 5 | 5 | 3
hour*nanograms/milliliter | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

22. Primary Outcome: AUC(0-inf) of GSK1278863 (Part B)
Description: as for outcome 21
Time Frame: Pre-dose and 2 hrs on Day 1 and 7; pre-dose, 1, 2,4, 8, 12 and 24 hrs post-dose on Day 14
Population: PK Population
Measure: Mean (Standard Deviation); unit: hour*nanograms/milliliter
Arm/Group | R1r (Cohort 5)
Number analyzed (Participants) | 26
hour*nanograms/milliliter | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

23. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Within a Participant Across All Treatments [AUC(0-t)] of GSK1278863 (Part A)
Description: The pharmacokinetic parameters were calculated by standard non-compartmental analysis according to current working practices and using WinNonlin Version 5.2 or higher. All calculations of non-compartmental parameters were based on actual sampling times. AUC (0-t) could not be determined as data was below the limit of quantification.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72 hrs post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: hour*nanograms/milliliter
Arm/Group | A/B (Cohort 1) | C/C (Cohort 2) | D (Cohort 3) | E/E (Cohort 4)
Number analyzed (Participants) | 9 | 5 | 5 | 3
hour*nanograms/milliliter | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification. | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

24. Primary Outcome: AUC(0-t) of GSK1278863 (Part B)
Description: as for outcome 23
Time Frame: Pre-dose and 2 hrs on Day 1 and 7; pre-dose, 1, 2,4, 8, 12 and 24 hrs post-dose on Day 14
Population: PK Population
Measure: Mean (Standard Deviation); unit: hour*nanograms/milliliter
Arm/Group | R1r (Cohort 5)
Number analyzed (Participants) | 26
hour*nanograms/milliliter | NA (NA) — NA indicates that data could not be determined as the data was below limit of quantification.

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected from start of study treatment through the final follow-up visit each of Part A {up to a maximum of 75 days (start of study treatment through final follow up 2 [28-32 days post last dose])} and B {up to a maximum of 53 days (start of study treatment through final follow up 2 [28-32 days post last dose])}
Description: All Subject Population was used to assess AEs and SAEs
Arm/Group | Placebo HVT (Cohort 1) | A/B (Cohort 1) | Placebo DFU SD (Cohort 2, 3, 4) | C (Cohort 2) | D (Cohort 3) | E (Cohort 4) | Placebo DFU RD (Cohort 5) | R1r (Cohort 5) | Sr (Cohort 5)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9 | 0/3 | 0/5 | 0/5 | 0/3 | 0/4 | 0/26 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9 | 0/3 | 0/5 | 0/5 | 1/3 | 1/4 | 0/26 | 1/4
Other Adverse Events (participants affected / at risk) | 1/4 | 2/9 | 1/3 | 0/5 | 0/5 | 1/3 | 1/4 | 0/26 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo HVT (Cohort 1) (N=4) | A/B (Cohort 1) (N=9) | Placebo DFU SD (Cohort 2, 3, 4) (N=3) | C (Cohort 2) (N=5) | D (Cohort 3) (N=5) | E (Cohort 4) (N=3) | Placebo DFU RD (Cohort 5) (N=4) | R1r (Cohort 5) (N=26) | Sr (Cohort 5) (N=4)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo HVT (Cohort 1) (N=4) | A/B (Cohort 1) (N=9) | Placebo DFU SD (Cohort 2, 3, 4) (N=3) | C (Cohort 2) (N=5) | D (Cohort 3) (N=5) | E (Cohort 4) (N=3) | Placebo DFU RD (Cohort 5) (N=4) | R1r (Cohort 5) (N=26) | Sr (Cohort 5) (N=4)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-07-31): https://cdn.clinicaltrials.gov/large-docs/04/NCT01831804/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT01831804/SAP_001.pdf